CLINICAL TRIAL: NCT00645710
Title: A Phase I/II Trial of Radioimmunotherapy (Y-90 cT84.66), Gemcitabine and Hepatic Arterial Infusion of Fudr for Metastatic Colorectal Carcinoma to the Liver
Brief Title: Hepatic Arterial Infusion of Floxuridine, Gemcitabine Hydrochloride, and Radiolabeled Monoclonal Antibody Therapy in Treating Liver Metastases in Patients With Metastatic Colorectal Cancer Previously Treated With Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04122; NCI-2010-01229; CDR0000590335 (Registry Identifier: PDQ)
Record Dates: First submitted 2008-03-27; First posted 2008-03-28 (Estimated); Results first posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-02

CONDITIONS: Liver Metastases; Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage IV Colon Cancer; Stage IV Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Gemcitabine; Floxuridine; Chromatography, Liquid; Mass Spectrometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive floxuridine as a continuous hepatic arterial infusion on days 1-14 and gemcitabine hydrochloride IV over 30 minutes on days 9 and 11. Patients also receive yttrium Y 90 anti-CEA monoclonal antibody cT84.66 IV over 25 minutes on day 9. Treatment repeats every 6 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Patients may receive an additional course of floxuridine in combination with systemic therapy at the discretion of the treating physician.
  Interventions: Drug: gemcitabine hydrochloride; Drug: floxuridine; Genetic: proteomic profiling; Other: matrix-assisted laser desorption/ionization time of flight mass spectrometry; Other: liquid chromatography; Radiation: yttrium Y 90 anti-CEA monoclonal antibody cT84.66; Other: laboratory biomarker analysis; Other: mass spectrometry; Other: pharmacological study

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; dFdCyd; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar; LY-188011
Drug: floxuridine — Given via hepatic arterial infusion
  Other Names: 5-FUDR; FdUrD; floxuridin; fluorodeoxyuridine; fluoruridine deoxyribose; FUdR
Genetic: proteomic profiling — Correlative studies
Other: matrix-assisted laser desorption/ionization time of flight mass spectrometry — Correlative studies
  Other Names: MALDI-TOF Mass Spectrometry
Other: liquid chromatography — Correlative studies
  Other Names: LC
Radiation: yttrium Y 90 anti-CEA monoclonal antibody cT84.66 — Given IV
Other: laboratory biomarker analysis — Correlative studies
Other: mass spectrometry — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as floxuridine and gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Hepatic arterial infusion uses a catheter to carry cancer-killing substances directly into the liver. Radiolabeled monoclonal antibodies can find tumor cells and carry tumor-killing substances to them without harming normal cells. Giving hepatic arterial infusion of floxuridine together with gemcitabine hydrochloride and radiolabeled monoclonal antibody therapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase I/II trial is studying the side effects and best dose of floxuridine when given as a hepatic arterial infusion together with gemcitabine hydrochloride and radiolabeled monoclonal antibody therapy and to see how well it works in treating liver metastases in patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and associated toxicities of concurrent hepatic arterial infusion (HAI) fluorodeoxypyrimidine (FUdR)/Decadron and intravenous gemcitabine combined with intravenous yttrium-90 (^90Y) chimeric T84.66 (cT84.66) in colorectal cancer patients after hepatic resection or maximum surgical debulking (to < 3 cm) of liver metastases.

II. To study the feasibility and toxicities of such adjuvant therapy following resection and/or ablation of liver metastases.

III. To evaluate the biodistribution, clearance and metabolism of ^90Y and ^111In (indium-iii) chimeric T84.66 administered intravenously.

IV. To estimate radiation doses to whole body, normal organs, and tumor through serial nuclear imaging.

V. To correlate proteomic profiles pre and post-therapy with toxicities and anti-tumor effects.

OUTLINE: This is a phase I, dose-escalation study of floxuridine followed by a phase II study.

Patients receive floxuridine as a continuous hepatic arterial infusion on days 1-14 and gemcitabine hydrochloride IV over 30 minutes on days 9 and 11. Patients also receive yttrium Y 90 anti-CEA monoclonal antibody cT84.66 IV over 25 minutes on day 9. Treatment repeats every 6 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.

Patients may receive an additional course of floxuridine in combination with systemic therapy at the discretion of the treating physician.

After completion of study treatment, patients are followed up at 3 and 6 months.

ELIGIBILITY:
Inclusion

* Patients must have a Karnofsky performance status of >= 60%; this must be met pre-surgery and pre-study therapy
* Patients must have histological confirmation of colorectal carcinoma and present with potentially resectable or abatable metachronous or synchronous hepatic metastases
* Patients must have colorectal tumors that produce CEA as documented by either immunohistochemistry or by an elevated serum CEA
* Prior radiotherapy, immunotherapy, or chemotherapy must have been completed at least four weeks prior to start of FUdR/RIT therapy on this study (6 weeks if mitomycin-C or nitrosoureas were part of last therapy) and patients must have recovered from all expected side effects of the prior therapy
* Laboratory values must be met pre-surgery and pre-study therapy
* Hemoglobin > 10 gm % (patients may be transfused to reach a hemoglobin > 10 gm %)
* WBC > 4000/ul
* Absolute granulocyte count of > 1,500/mm^3
* Platelets > 150,000/ul
* Patients may have history of prior malignancy for which the patient has been disease-free for five years with the exception of basal or squamous cell skin cancers or carcinoma in situ of the cervix
* Patients must have no prior history of radiation therapy to the liver
* Total bilirubin < 1.5 (unless reversibly obstructed due to the metastatic tumor)
* Serum creatinine of < 2.0
* Patients must have evidence of intrahepatic metastases involving < 60% of the functioning liver
* Patients cannot have evidence of extrahepatic disease with the following exceptions: patients known to have a resectable "anastomotic" or local recurrence of their tumor; patients who undergoing their initial surgery for resection of their primary colorectal carcinoma can have potentially resectable porta hepatis and/or mesenteric lymph node involvement in addition to liver metastases; patients who have disease extension from the liver metastasis that can be resected en bloc (e.g., diaphragm, kidney, and abdominal wall); patients who have minimal, potentially resectable to less than 3 cm extrahepatic disease
* The pre-operative eligibility checklist must be completed
* If a patient has previously received murine or chimeric antibody, then serum anti-antibody testing must be negative (This must be met pre-surgery if possible)
* Serum HIV testing and hepatitis B surface antigen and C antibody testing must be negative
* Women of childbearing potential must have a negative serum pregnancy test prior to entry and while on study must be practicing an effective form of contraception (This must be met pre-surgery and pre-study therapy)
* Patients must have resectable or abatable liver metastases as determined by the attending surgeon
* Colorectal carcinoma must be confined to the liver except as noted above
* Patients with limited extrahepatic disease as defined (primary, lymph node, or anastomotic recurrence) must have disease resected or debulked to less than 3 cm in greatest dimension
* To receive study therapy, patients must be at least 3 weeks post-surgery but no more than 16 weeks post surgery and without evidence of post-operative complications, such as infection or poor wound healing
* Patients must have < 40% liver resected at the close of completion of the hepatic resection

Exclusion

* Patients that have received radiation therapy to greater than 50% of their bone marrow
* Patients with any nonmalignant intercurrent illness (example cardiovascular, pulmonary, or central nervous system disease) which is either poorly controlled with currently available treatment or which is of such severity that the investigators deem it unwise to enter the patient on protocol shall be ineligible
* Biopsy-proven chronic active hepatitis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-02-11; Primary Completion 2018-02-07 (Actual); Study Completion 2018-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Wong, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1- FUdR 0.10 mg/kg/Day: Patients receive floxuridine as a continuous hepatic arterial infusion on days 1-14 (dose level 0.10 mg/kg/day) and gemcitabine hydrochloride IV (105 mg/m^2) over 30 minutes on days 9 and 11. Patients also receive yttrium Y 90 anti-CEA monoclonal antibody cT84.66 IV (16.6 mCi/m^2) over 25 minutes on day 9. Treatment repeats every 6 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Patients may receive an additional course of floxuridine in combination with systemic therapy at the discretion of the treating physician.
- Dose Level 2 - FUdR 0.15 mg/kg/Day: Patients receive floxuridine as a continuous hepatic arterial infusion on days 1-14 (dose level 0.15 mg/kg/day) and gemcitabine hydrochloride IV (105 mg/m^2) over 30 minutes on days 9 and 11. Patients also receive yttrium Y 90 anti-CEA monoclonal antibody cT84.66 IV (16.6 mCi/m^2) over 25 minutes on day 9. Treatment repeats every 6 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Patients may receive an additional course of floxuridine in combination with systemic therapy at the discretion of the treating physician.
- Dose Level 3 - FUdR 0.20 mg/kg/Day: Patients receive floxuridine as a continuous hepatic arterial infusion on days 1-14 (dose level 0.20 mg/kg/day) and gemcitabine hydrochloride IV (105 mg/m^2) over 30 minutes on days 9 and 11. Patients also receive yttrium Y 90 anti-CEA monoclonal antibody cT84.66 IV (16.6 mCi/m^2) over 25 minutes on day 9. Treatment repeats every 6 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Patients may receive an additional course of floxuridine in combination with systemic therapy at the discretion of the treating physician.
Period: Overall Study
Arm/Group | Dose Level 1- FUdR 0.10 mg/kg/Day | Dose Level 2 - FUdR 0.15 mg/kg/Day | Dose Level 3 - FUdR 0.20 mg/kg/Day
Started | 3 | 3 | 10
Completed | 3 | 3 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 1 - FUdR 0.10 mg/kg/Day: Patients receive floxuridine as a continuous hepatic arterial infusion on days 1-14 (starting dose level 0.10 mg/kg/day) and gemcitabine hydrochloride IV (105 mg/m^2) over 30 minutes on days 9 and 11. Patients also receive yttrium Y 90 anti-CEA monoclonal antibody cT84.66 IV (16.6 mCi/m^2) over 25 minutes on day 9. Treatment repeats every 6 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Patients may receive an additional course of floxuridine in combination with systemic therapy at the discretion of the treating physician.
- Dose Level 2 - FUdR 0.15 mg/kg/Day: Patients receive floxuridine as a continuous hepatic arterial infusion on days 1-14 (starting dose level 0.15 mg/kg/day) and gemcitabine hydrochloride IV (105 mg/m^2) over 30 minutes on days 9 and 11. Patients also receive yttrium Y 90 anti-CEA monoclonal antibody cT84.66 IV (16.6 mCi/m^2) over 25 minutes on day 9. Treatment repeats every 6 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Patients may receive an additional course of floxuridine in combination with systemic therapy at the discretion of the treating physician.
- Dose Level 3 - FUdR 0.20 mg/kg/Day: Patients receive floxuridine as a continuous hepatic arterial infusion on days 1-14 (starting dose level 0.20 mg/kg/day) and gemcitabine hydrochloride IV (105 mg/m^2) over 30 minutes on days 9 and 11. Patients also receive yttrium Y 90 anti-CEA monoclonal antibody cT84.66 IV (16.6 mCi/m^2) over 25 minutes on day 9. Treatment repeats every 6 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Patients may receive an additional course of floxuridine in combination with systemic therapy at the discretion of the treating physician.
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 - FUdR 0.10 mg/kg/Day | Dose Level 2 - FUdR 0.15 mg/kg/Day | Dose Level 3 - FUdR 0.20 mg/kg/Day | Total
Number analyzed (Participants) | 3 | 3 | 10 | 16
Age, Continuous [Median (Full Range); unit: years] | 60 [50 to 66] | 54 [45 to 77] | 53 [35 to 66] | 56 [35 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3 | 6
  Male | 2 | 1 | 7 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 2 | 3
  Hispanic | 1 | 0 | 2 | 3
  Caucasian | 2 | 2 | 5 | 9
  Unknown | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 10 | 16
Karnofsky Performance Status for Assessment of Functional Impairment [Median (Full Range); unit: units on a scale] — 100 - Normal no complaints. 90 - Able to carry on normal activity; minor signs or symptoms of disease.80 - Normal activity with effort. 70 - Cares for self; unable to carry on normal activity or active work. 60 - Requires occasional assistance, but is able to care for most personal needs. 50 - Requires considerable assistance and frequent medical care. 40 - Disabled; requires special care and assistance. 30 - Severely disabled; hospitalization indicated although death not imminent. 20 - Very sick. Hospitalization necessary. Active supportive treatment necessary.10 - Moribund. 0 - Dead.
  units on a scale | 90 [80 to 90] | 90 [90 to 90] | 90 [60 to 100] | 90 [60 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Dose Limiting Toxicity
Description: Dose Limiting Toxicity (DLT) defined as any treatment-related grade grade 3 nonhematologic toxicity not reversible to grade 2 or less within 24 hours, or any grade 4 toxicity.Up to three cycles of therapy were allowed with DLTs determined based on first cycle tolerance. Toxicity was graded using the National Cancer Institute Common Toxicity Criteria version 2.0.
Time Frame: 4 weeks from start of treatment, up to 2 years.
Population: All patients receiving treatment were evaluated for DLT.
Measure: Number; unit: participants with DLTs
Arm/Group | Dose Level 1- FUdR 0.10 mg/kg/Day | Dose Level 2 - FUdR 0.15 mg/kg/Day | Dose Level 3 - FUdR 0.20 mg/kg/Day
Number analyzed (Participants) | 3 | 3 | 10
participants with DLTs | 0 | 0 | 1

2. Primary Outcome: Recommended Phase II Dose
Description: The maximum tolerated dose (MTD) of HAI FUdR in combination with intravenous gemcitabine and 90Y-DTPA-cT84.66 is based on toxicities observed during the first cycle and is defined as the highest dose tested in which fewer than 33% of patients experience an attributable DLT to the study drug, when at least 6 patients are treated at that dose and are evaluable for toxicity. Dose escalations proceeded according to a standard 3+3 design.
Time Frame: 4 weeks from start of treatment, up to 2 years.
Population: All patients observed for 56 days while receiving a full course of therapy or who experienced a DLT. Patients withdrawing before completion of the first course, for reasons other than DLT, were replaced.
Measure: Number; unit: mg/kg/day
Groups:
- RIT/Gemcitabine/FUdR: Patients receive floxuridine as a continuous hepatic arterial infusion on days 1-14 (starting dose level 0.10 mg/kg/day) and gemcitabine hydrochloride IV (105 mg/m^2) over 30 minutes on days 9 and 11. Patients also receive yttrium Y 90 anti-CEA monoclonal antibody cT84.66 IV (16.6 mCi/m^2) over 25 minutes on day 9. Treatment repeats every 6 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Patients may receive an additional course of floxuridine in combination with systemic therapy at the discretion of the treating physician.
Arm/Group | RIT/Gemcitabine/FUdR
Number analyzed (Participants) | 10
mg/kg/day | 0.20

3. Secondary Outcome: Overall Survival
Description: Estimated using the product-limit method of Kaplan and Meier. Event defined as death due to any cause.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose Level 1- FUdR 0.10 mg/kg/Day | Dose Level 2 - FUdR 0.15 mg/kg/Day | Dose Level 3 - FUdR 0.20 mg/kg/Day
Number analyzed (Participants) | 3 | 3 | 10
Months | 23.2 [18.9 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 73.2 [27.4 to 132.9] | 41.2 [18.4 to 65.5]

4. Secondary Outcome: Progression-free Survival
Description: Estimated using the product-limit method of Kaplan and Meier. Progression is defined as a 25% increase in the sum of products of measurable lesions over the smallest sum observed, or appearance of any lesions that had disappeared, or appearance of any new lesion/site.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose Level 1- FUdR 0.10 mg/kg/Day | Dose Level 2 - FUdR 0.15 mg/kg/Day | Dose Level 3 - FUdR 0.20 mg/kg/Day
Number analyzed (Participants) | 3 | 3 | 10
Months | 8.3 [5.0 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 11.5 [6.6 to 12.9] | 9.6 [1.0 to 19.0]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 6 years and 11 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Groups:
- Dose Level 1- FUdR 0.10 mg/kg/Day: Patients receive floxuridine as a continuous hepatic arterial infusion on days 1-14 (starting dose level 0.10 mg/kg/day) and gemcitabine hydrochloride IV (105 mg/m^2) over 30 minutes on days 9 and 11. Patients also receive yttrium Y 90 anti-CEA monoclonal antibody cT84.66 IV (16.6 mCi/m^2) over 25 minutes on day 9. Treatment repeats every 6 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Patients may receive an additional course of floxuridine in combination with systemic therapy at the discretion of the treating physician.
- Dose Level 2- FUdR 0.15 mg/kg/Day: Patients receive floxuridine as a continuous hepatic arterial infusion on days 1-14 (starting dose level 0.15 mg/kg/day) and gemcitabine hydrochloride IV (105 mg/m^2) over 30 minutes on days 9 and 11. Patients also receive yttrium Y 90 anti-CEA monoclonal antibody cT84.66 IV (16.6 mCi/m^2) over 25 minutes on day 9. Treatment repeats every 6 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Patients may receive an additional course of floxuridine in combination with systemic therapy at the discretion of the treating physician.
- Dose Level 3- FUdR 0.20 mg/kg/Day: Patients receive floxuridine as a continuous hepatic arterial infusion on days 1-14 (starting dose level 0.20 mg/kg/day) and gemcitabine hydrochloride IV (105 mg/m^2) over 30 minutes on days 9 and 11. Patients also receive yttrium Y 90 anti-CEA monoclonal antibody cT84.66 IV (16.6 mCi/m^2) over 25 minutes on day 9. Treatment repeats every 6 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Patients may receive an additional course of floxuridine in combination with systemic therapy at the discretion of the treating physician.
Arm/Group | Dose Level 1- FUdR 0.10 mg/kg/Day | Dose Level 2- FUdR 0.15 mg/kg/Day | Dose Level 3- FUdR 0.20 mg/kg/Day
All-Cause Mortality (participants affected / at risk) | 2/3 | 3/3 | 8/10
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 2/10
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1- FUdR 0.10 mg/kg/Day (N=3) | Dose Level 2- FUdR 0.15 mg/kg/Day (N=3) | Dose Level 3- FUdR 0.20 mg/kg/Day (N=10)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1- FUdR 0.10 mg/kg/Day (N=3) | Dose Level 2- FUdR 0.15 mg/kg/Day (N=3) | Dose Level 3- FUdR 0.20 mg/kg/Day (N=10)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (3) | 2 (4) | 9 (16)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Premature ventricular contractions (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 2 (3) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (4)
Anal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3) | 2 (2) | 3 (5)
Diarrhea (Gastrointestinal disorders) | 3 (4) | 2 (4) | 7 (11)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (3)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (8) | 3 (4) | 7 (13)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 4 (5)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 2 (2) | 2 (3) | 1 (1)
Disease progression (General disorders) | 1 (1) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 3 (9) | 3 (11) | 10 (25)
Fever (General disorders) | 2 (3) | 2 (3) | 2 (2)
Localized edema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 1 (2) | 6 (8)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (3)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (11) | 3 (9) | 10 (21)
Alkaline phosphatase increased (Investigations) | 2 (5) | 2 (4) | 7 (15)
Aspartate aminotransferase increased (Investigations) | 3 (11) | 3 (12) | 9 (22)
Bilirubin increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Haptoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinemia (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolemia (Investigations) | 1 (1) | 3 (4) | 1 (1)
Leukocyte count decreased (Investigations) | 1 (2) | 0 (0) | 9 (19)
Leukopenia (Investigations) | 3 (8) | 3 (9) | 2 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 9 (13)
Lymphopenia (Investigations) | 3 (5) | 3 (11) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (6) | 2 (6) | 10 (16)
Platelet count decreased (Investigations) | 2 (5) | 2 (8) | 7 (14)
Serum cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Weight gain (Investigations) | 1 (1) | 3 (3) | 3 (6)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 5 (6)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (12)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3) | 2 (6) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (3) | 2 (2) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (3) | 1 (2) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (6) | 1 (4)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (3)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum triglycerides increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 5 (8)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (5) | 2 (4) | 6 (8)
Taste alteration (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (3)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Bladder pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal hemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 4 (4)
Skin disorder (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Flushing (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Hemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (3)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT00645710/Prot_SAP_000.pdf